CLINICAL TRIAL: NCT07336043
Title: Optimizing Regional Analgesia in Pediatric Laparoscopic Splenectomy: External Oblique Intercostal Block Versus Transversus Abdominis Plane Block: Randomized Controlled Study
Brief Title: External Oblique Intercostal Block Versus Transversus Abdominis Plane Block in Pediatric Laparoscopic Splenectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Esraa Rabie Amer, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR131092/11/25
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Regional Block; Pediatric; Laparoscopic Splenectomy; External Oblique Intercostal Block; Transversus Abdominis Plane Block
Keywords: Pediatric; External Oblique Intercostal Block; Transversus Abdominis Plane Block; Regional Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOI group (Group E) (Experimental): 30 patients will receive ultrasound-guided left EOI block
  Interventions: Procedure: EOI group
- TAP group (Group T) (Experimental): 30 patients will receive ultrasound-guided left TAP block
  Interventions: Procedure: TAP group

INTERVENTIONS:
Procedure: EOI group — patients will receive ultrasound-guided left EOI block.
  Arms: EOI group (Group E)
Procedure: TAP group — patients will receive ultrasound-guided left TAP block
  Arms: TAP group (Group T)

SUMMARY:
The aim of study is to compare the efficacy of the External Oblique Intercostal plane block with the Transversus Abdominis Plane block in acute postoperative pain control in pediatric patients undergoing laparoscopic Splenectomy.

DETAILED DESCRIPTION:
Optimal postoperative pain control in children is particularly challenging despite advances in multimodal pharmaceutical strategies. Laparoscopic approaches have improved postoperative outcomes when compared to open surgery, particularly in terms of postoperative pain. Pain after laparoscopic surgeries has three components; including incisional, visceral, and referred shoulder pain secondary to peritoneal insufflation. Opioid analgesia can be an effective adjunct to an existing non-opioid pain regimen. However, opioids are known to decrease bowel motility, result in nausea, and cause respiratory depression, particularly in the pediatrics. Traditionally, neuraxial blocks have been used for abdominal surgeries but in patients with low platelet count as splenectomy, this might not be a feasible option.

Effective fascial plane blocks have recently become popular as candidates to be a part of multimodal analgesia, especially for patients who require limited use of drugs in multimodal analgesia (such as liver failure, renal failure, platelet dysfunction, and peptic ulcer) or those with hypersensitivity to any of these drugs. As there are potential advantages such as a longer distance between the needle and neurovascular structures, less motor blockade and less hemodynamic change, fascial plane blocks can provide effective solutions to many difficulties faced by anesthesiologists in the perioperative period. Transversus Abdominis Plane block has emerged as an effective method to minimize postoperative pain in adult patients undergoing abdominal surgery. Several randomized trials in children undergoing laparoscopic appendicectomy, minimally invasive cholecystectomy, and other laparoscopic abdominal procedures have demonstrated that ultrasound-guided Transversus Abdominis Plane block reduces pain scores, opioid consumption, and even pulmonary complications such as atelectasis when compared with port site infiltration or systemic analgesia alone.

External oblique intercostal block is a novel block, which has been described as an important modification of the fascial plane blocks that can consistently involve the upper lateral abdominal walls. External oblique intercostal block block targets the external oblique intercostal plane, allowing for effective analgesia across the upper abdominal wall, including both median and lateral regions. This contrasts with the Transversus Abdominis Plane block block, which may not adequately cover the lateral cutaneous intercostal branches, limiting its effectiveness in certain surgical procedures. Many previous studies that have concentrated on the use of different TAP block strategies, including subcostal Transversus Abdominis Plane block; have shown that it could not sufficiently block the lateral cutaneous intercostal branches.

The aim of study is to compare the efficacy of the External Oblique Intercostal plane block with the Transversus Abdominis Plane block in acute postoperative pain control in pediatric patients undergoing laparoscopic Splenectomy.

* Primary outcome: Postoperative Numerical rating scale score.
* Secondary outcomes

  1. The amount of morphine consumption postoperatively.
  2. Time to first opioid request .
  3. Intraoperative fentanyl consumption.
  4. Intraoperative vital signs including mean arterial pressure and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Children of both gender,
* aged 8 to 16 years with American Society of Anesthesiologists Physical Status I to III,
* who were scheduled for laparoscopic Splenectomy surgery.

Exclusion Criteria:

* Parents declined to participate in the trial.
* Physical or developmental delay.
* Pre-existing renal or cardiovascular disease, bone disease, or gastrointestinal disorders.
* Infection at proposed injection sites.
* Prior major abdominal surgery

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale score | Numerical rating scale score will be assessed postoperatively 10, 30 and 60 minutes then 2 , 4 , 6 , 12 , 24 hours postoperatively
  Numerical rating scale score

SECONDARY OUTCOMES:
Intraoperative Heart rate values | every 15 minutes until end of surgery
  Intraoperative Heart rate values at the time of port placement and every 15 min until end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be provided if it was needed
Supporting Information: Study Protocol, SAP, ICF